CLINICAL TRIAL: NCT00466011
Title: Validation of the Stardust Cardio-Respiratory Recorder
Acronym: Stardust
Status: Completed | Type: Observational
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Lia Azeredo-Bittencourt, Prof. Dr., Associação Fundo de Incentivo à Pesquisa
Other Study IDs: 0099/07
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Introduction: The full night polysomnography (PSG) in sleep lab is the gold standard to Obstructive Sleep Apnea (OSA) diagnosis. However, there is a need to evaluate simple and accurate home diagnostic equipment that can reliably detect or exclude OSA. The aim of our study was to evaluate if an ambulatory portable monitor (SD) is accurate to measure apnea-hypopnea index (AHI) in OSA patients referred to a Sleep Lab. Methods: Patients with clinical suspicion of OSA were selected. Three-order randomized evaluations had been performed within a period of two weeks: the 1) SD (Stardust®, Respironics, Inc, USA) was used at patients home (SD home), 2) SD was used simultaneously with PSG in the sleep lab (SD+PSG lab) and 3) PSG was performed without the use of SD (PSG lab). Four AHI were generated and analyzed: AHI from SD home, AHI from SD of SD+PSG lab, AHI from PSG of PSG+SD lab and AHI from PSG lab. The analyses of SDs and PSGs recordings were performed by two blinded technicians.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to Sleep Disorder Center because of:

  * Excessive daytime sleepiness,
  * Loud snoring,
  * Witnessed apnea.
* Patient with ability to provide consent, ability and willingness to follow study procedures.

Exclusion Criteria:

* Suspicion of insomnia,
* Restless leg syndrome,
* Periodic limb movements; or
* Other non-OSA sleep disorders.
* Patient experiencing acute illness, patients who are medically complex, and patients requiring supplemental oxygen or mechanical ventilation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients with complains of OSA
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Tufik, MD, PhD, Study Director — Associacao Fundo de Incentivo a Psicofarmcologia
Locations (1):
- AFIP, São Paulo, São Paulo, Brazil